CLINICAL TRIAL: NCT05727423
Title: Safety and Efficacy of Dapagliflozin in the Treatment of Heart Failure in Non-diabetic Egyptian Patients
Brief Title: Dapagliflozin in the Treatment of Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Madonna salama hanna, Teaching Assistant, Helwan University
Other Study IDs: 05H2021
Record Dates: First submitted 2023-02-05; First posted 2023-02-14 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
prospectively evaluation the safety and efficacy of the Sodium-glucose Cotransporter-2 (SGLT2) inhibitor dapagliflozin in non-diabetic patients with heart failure and a reduced ejection fraction

DETAILED DESCRIPTION:
Heart failure (HF) is a complex clinical syndrome characterized by the reduced ability of the heart to pump and/or fill with blood. From a physiological point of view, HF can be defined as an inadequate cardiac output to meet metabolic demands.

HF is a growing public health problem, with an estimated 63 million people affected worldwide , with HF being the underlying cause of more than 1 million hospitalizations every year. These hospitalizations are associated with poor prognosis (50% rate of re-hospitalization within 6 months after discharge and around 33% rate of death within 12 months after discharge), In addition, the prevalence of patient with HF and reduced ejection fraction (HFrEF) is higher and has greater mortality rates than those with preserved ejection fraction (HFpEF).

Sodium-glucose Cotransporter-2(SGLT2) inhibitors are a novel class of anti diabetic agents that promote urinary glucose excretion by inhibiting glucose and sodium reabsorption from the renal proximal tubules and have recently been investigated in several large randomized controlled trials for cardiovascular safety and efficacy in patients with type 2 diabetes .

More recently, the DAPA-HF trial which showed that dapagliflozin significantly improved the outcomes of patients with HFrEF and reduced the risk of the composite outcome of CV death or the worsening of HF versus placebo by 26% irrespective of the presence or absence of T2DM, demonstrated the significance of SGLT2 inhibitors as novel therapeutic agents in heart failure.

In May 2020,The FDA approved AstraZeneca's dapagliflozin (Forxiga) for the treatment of heart failure with reduced ejection fraction (HFrEF) in adults with and without type 2 diabetes (T2D), marking the first time a drug in a class developed for diabetes was approved for heart failure even if diabetes is not present.

This study is established to investigate safety and efficacy of dapagliflozin in non-diabetic patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* patients age > 18 years
* Diagnosis of heart failure NYHA class II- IV
* LVEF ≤ 40% on echocardiography

Exclusion Criteria:

* Estimated glomerular filtration rate <30 ml/min/1.73m2

  * Pregnant or lactating women

Ages: 19 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In the cardiology department at Ain Shams university hospitals, stable heart failure patients with reduced ejection fraction should fulfill the inclusion and exclusion criteria mentioned above.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-01-28 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
left ventricular ejection fraction | 6 months
  Assessment of Echo parameters of LV-systolic function as EF

SECONDARY OUTCOMES:
left ventricular end-systolic volume, left ventricular end-diastolic volume | 6 months
  Assessment of Echo parameters of LV-systolic function as LVESV, LVEDV
E/e', LAVI, septal e' | 6 months
  Assessment of Echo parameters of LV- diastolic function as E/e', LAVI, septal e'

CONTACTS AND LOCATIONS:
Locations (1):
- cardiology department at Ain Shams university hospitals, Cairo, Egypt

REFERENCES:
- [Background] Coronel R, de Groot JR, van Lieshout JJ. Defining heart failure. Cardiovasc Res. 2001 Jun;50(3):419-22. doi: 10.1016/s0008-6363(01)00284-x. No abstract available. PMID 11376615
- [Background] Lam CSP, Gamble GD, Ling LH, Sim D, Leong KTG, Yeo PSD, Ong HY, Jaufeerally F, Ng TP, Cameron VA, Poppe K, Lund M, Devlin G, Troughton R, Richards AM, Doughty RN. Mortality associated with heart failure with preserved vs. reduced ejection fraction in a prospective international multi-ethnic cohort study. Eur Heart J. 2018 May 21;39(20):1770-1780. doi: 10.1093/eurheartj/ehy005. PMID 29390051
- [Background] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Background] Rahmoune H, Thompson PW, Ward JM, Smith CD, Hong G, Brown J. Glucose transporters in human renal proximal tubular cells isolated from the urine of patients with non-insulin-dependent diabetes. Diabetes. 2005 Dec;54(12):3427-34. doi: 10.2337/diabetes.54.12.3427. PMID 16306358